CLINICAL TRIAL: NCT01783600
Title: NanoCross BTK, a Prospective, Non-randomized, Multicenter, Controlled Trial Evaluating the Performance of the NanoCrossTM .014 Balloon Catheter in Infrapopliteal Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-111125
Record Dates: First submitted 2013-01-25; First posted 2013-02-05 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Infrapopliteal lesions; balloon catheter
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NanoCross .014 balloon catheter (Other): NanoCross .014 balloon catheter
  Interventions: Device: NanoCross .014 balloon catheter

INTERVENTIONS:
Device: NanoCross .014 balloon catheter

SUMMARY:
The objective of this clinical evaluation is to evaluate the immediate and long-term (up to 12 months) outcome of NanoCrossTM balloon catheter (Covidien) in a prospective, non-randomised, controlled investigation for the treatment of patients with critical limb ischemia (Rutherford 4-5) due to the presence of lesions of minimally 10cm in length at the level of the below-the-knee arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with rest pain or minor tissue loss (Rutherford class 4 or 5)
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient has a projected life-expectancy of at least 12 months
* Patient is eligible for treatment with the NanoCrossTM .014 balloon catheter (Covidien)
* Male, infertile female, or female of child bearing potential practicing an acceptable method of birth control with a negative pregnancy test within 7 days prior to study procedure
* De novo lesion or restenotic lesion after PTA in the infrapopliteal arteries,suitable for endovascular therapy
* Total target lesion length minimally 100mm
* Target vessel diameter visually estimated to be >1.5mm and <4.0mm
* Guidewire and delivery system successfully traversed lesion
* At least one non-occluded crural artery with angiographically documented run- off to the foot.

Exclusion Criteria:

* Patient refusing treatment
* The reference segment diameter is not suitable for the available balloon design
* Untreated flow-limiting inflow lesions
* Perioperative unsuccessful ipsilateral percutaneous vascular procedure to treat inflow disease just prior to enrollment
* Any previous surgery in the target vessel (including prior ipsilateral crural bypass)
* Aneurysm in the target vessel
* Target lesion has severe calcification as determined by physician's discretion
* Non-atherosclerotic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis)
* Severe medical comorbidities (untreated CAD/CHF, severe COPD, metastatic malignancy, dementia, etc) or other medical condition that would preclude compliance with the study protocol or 1-year life expectancy
* Major distal amputation (above the transmetatarsal) in the study limb or non- study limb
* Septicemia or bacteremia
* Any previously known coagulation disorder, including hypercoagulability
* Contraindication to anticoagulation or antiplatelet therapy
* Known allergy to contrast media that cannot be adequately pre-medicated prior to the study procedure
* Patient with known hypersensitivity to heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT) type II
* Currently participating in another clinical research trial
* Angiographic evidence of intra-arterial thrombus or atheroembolism from inflow treatment
* Target lesion access not performed by transfemoral approach.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
primary Patency | 12 Months
  Primary patency at 12 months, defined as absence of restenosis (≥50% stenosis) or occlusion within the originally treated lesion based on duplex ultrasound (systolic velocity ratio no greater than 2.4) and without prior TLR are defined as being primary patent at the 12-month follow-up

SECONDARY OUTCOMES:
Technical success | Day 0 (=procedure date)
  Technical success, defined as the ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30%.
Hemodynamic primary patency | 1 and 6 months follow-up
  Hemodynamic primary patency rate at 1 and 6-month follow-up. Patients that present without a hemodynamically significant stenosis at the target area on duplex ultrasound (systolic velocity ratio no greater than 2.4) and without prior TLR are defined as being primary patent at the given follow-up.
Limb-salvage rate | 1, 6 and 12 months follow-up
  Limb-salvage rate at all follow-up visits, defined as absence of major amputation. Major amputation is defined as amputation at or above the ankle, as opposed to minor amputation, being an amputation at or below metatarsal level, preserving functionality of the foot).
Primary assisted patency rate | 1, 6, 12-month follow-up
  Primary assisted patency rate at 1, 6, 12-month follow-up. Defined as flow through the treated lesion maintained by repeat percutaneous intervention completed prior to complete vessel closure.
Secondary patency rate | 1, 6, 12-month follow-up
  Secondary patency rate at 1, 6, 12-month follow-up. Defined as flow through the treated lesion maintained by repeat percutaneous intervention after occlusion of the target lesion.
Target lesion revascularization | 1 day, 1 month, 6 month and 12 month follow-up
  Target lesion revascularization (TLR) is defined as a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5 mm proximal and distal to the treated lesion edge.
Clinical success at follow-up | 1 day and 1, 6, 12-month follow-up
  Clinical success at follow-up is defined as an improvement of Rutherford classification at 1 day and 1, 6, 12-month follow-up of one class or more as compared to the pre-procedure Rutherford classification.
Number of patients with Serious Adverse Events (SAE) as a measure of safety | 1 day, 1 month, 6 month and 12 month follow-up
  Serious adverse events as defined as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - OLV Aalst, Alast
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - RZ Heilig Hart Tienen, Tienen